CLINICAL TRIAL: NCT05889845
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Candin for the Treatment of Common Warts (Verruca Vulgaris) in Adolescents and Adults
Brief Title: Candin for the Treatment of Common Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nielsen BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFW-3A
Record Dates: First submitted 2023-05-02; First posted 2023-06-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Common Warts (Verruca Vulgaris)
Keywords: Common wart; Intralesional injection; Candida albicans; Immunotherapy
MeSH Terms: conditions — Warts

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded site staff will prepare syringes of study drug for administration by blinded study staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Candin treatment (Experimental): Candida albicans Skin Test Antigen for Cellular Hypersensitivity will be administered as a 0.5 mL injection at the region of the interdigitated base of the treatment wart (epidermal/dermal junction) every 2 weeks for up to 10 injections
  Interventions: Drug: Candin, Intradermal Solution
- Placebo (Placebo Comparator): Matching placebo (sterile saline) will be administered as a 0.5 mL injection at the region of the interdigitated base of the treatment wart (epidermal/dermal junction) every 2 weeks for up to 10 injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candin, Intradermal Solution — Injection at the base of the selected wart
  Arms: Candin treatment
Drug: Placebo — Injection at the base of the selected wart
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare outcome in healthy subjects 12 years of age and older with at least 3, but no more than 20, common warts (Verruca vulgaris) following treatment with Candin or placebo. The main questions it aims to answer are:

* does treatment with Candin result in better clearance of warts than placebo
* how many injections are required to result in wart clearance Participants will
* have one wart selected for injection every two weeks until clearance
* return 12 weeks after wart clearance for assessment of durability of response

DETAILED DESCRIPTION:
This study involves a comparison of an equal volume injection of Candin with an injection of placebo (unpreserved normal saline solution) in common warts. Subjects will be randomized 2:1 to receive Candin or placebo. During the Treatment Period, 1 dose (0.5 mL) of investigational product (IP) will be injected every 2 weeks into a single treatment wart until either clinical clearance of the treatment wart is achieved or a total of 10 injections have been administered.

Subjects achieving clinical clearance of the treatment wart will receive a final injection at the site of the cleared wart and then immediately enter the Observational Period for 12 weeks. Complete resolution is achieved when a subject demonstrates clinical clearance for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 3, but not more than 20 common warts (Verruca vulgaris)
* Willing to agree to use adequate contraception methods during the study

Exclusion Criteria:

* Systemic or localized diseases, conditions, or medications that could interfere with the assessment of safety or efficacy or that compromise immune function
* Candin delayed type hypersensitivity reaction test wheal sized < 5 mm or > 25 mm at the Baseline Visit
* History of keloid formation
* Prior treatment of common warts with liquid nitrogen, carbon dioxide, electrodesiccation, laser, surgery, salicylic acid, etc., that, in the Investigator's opinion, does not exhibit complete healing from the treatment
* Treatment with immunotherapy (e.g., diphenylcyclopropenone [DPCP], dinitrochlorobenzene [DNCB], or other), imiquimod, 5-fluorouracil, bleomycin, or podophyllin within 12 weeks of the Baseline Visit or during the study
* Prior treatment with Candida albicans within 12 weeks of the Baseline Visit or during the study
* Systemic treatment with an immunosuppressive drug during the study or in the 6 months or 5 half lives prior to the Baseline Visit or during the study (e.g., azathioprine, 6 mercaptopurine, methotrexate, infliximab, adalimumab, etanercept, systemic steroids [topical or inhaled steroids are acceptable]).
* Use of cantharidin or an investigational agent or device within the 30 days prior to the Baseline Visit or during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete resolution of the treatment wart | Twelve weeks after last injection
  Absence of visual or measurable wart maintained through the entire Observational Period for injected wart

SECONDARY OUTCOMES:
Time to wart clearance | Up to 27 weeks
  Time from first injection to achieving clinical clearance of the treatment wart. Clinical clearance is no evidence of the wart by visual inspection.
Number of participants with clinical clearance of at least 50% of all measured warts | Up to 27 weeks
  The injected wart and up to five other warts will be measured. Clinical clearance is no evidence of the wart by visual inspection.
Number of participants with clinical clearance of all measured warts | Up to 27 weeks
  The injected wart and up to five other warts will be measured. Clinical clearance is no evidence of the wart by visual inspection.
Time to clinical clearance of all measured warts | Up to 27 weeks
  The injected wart and up to five other warts will be measured. Clinical clearance is no evidence of the wart by visual inspection.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Cahaba Dermatology, Birmingham, Alabama
  - Arkansas Pediatric Clinic, Bryant, Arkansas
  - Johnson Dermatology, Fort Smith, Arkansas
  - Dermatology Clinic of Arkansas, Hot Springs, Arkansas
  - Velocity Clinical La Mesa, La Mesa, California
  - Long Beach Research, Long Beach, California
  - Integrative Skin Research, Sacramento, California
  - Velocity Clinical Englewood, Englewood, Colorado
  - Kaminska Dermatology, Chicago, Illinois
  - Integrated Dermatology of Newton-Brighton, Brighton, Massachusetts
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Schlessinger MD, Omaha, Nebraska
  - Advocare Berlin Medical Associates, Berlin, New Jersey
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Velocity Clinical Spartanburg, Spartanburg, South Carolina
  - DermResearch, Austin, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Velocity Clinical Hampton, Hampton, Virginia

IPD SHARING:
Plan to Share IPD: No